CLINICAL TRIAL: NCT05766280
Title: Internet Assisted Career-Oriented Soft-skills Training (iCareer) for Transition Age Youth with Mental Health Conditions: a Randomized Controlled Trial
Brief Title: Internet Assisted Career-Oriented Soft-skills Training for Transition Age Youth with Mental Health Conditions
Acronym: iCareer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Weili Lu, Ph.D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2022001761; 90IFRE0071 (Other Grant/Funding Number: DHHS: Administration for Community Living)
Record Dates: First submitted 2023-02-16; First posted 2023-03-13 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Mental Health Wellness 1; Mental Health Wellness 2; Occupational Problems
Keywords: transition age youth; mental health conditions; employment
MeSH Terms: interventions — Employment

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Assessors will not be providing the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Soft Skills Training Intervention via telehealth
  Interventions: Behavioral: iCareer Soft Skills Training for Employment
- Control (No Intervention): Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: iCareer Soft Skills Training for Employment — The telehealth iCareer intervention will be delivered during regular educational or vocational services (i.e., services from the Office of Disability Services (ODS) and/or from the school or college counseling center). Six modules of Soft Skills Training (SST), four group sessions for each module with 60 to 90 min for each session (depending on group size) will be delivered by trained project staff (graduate counseling student assistant or graduate counseling intern) via HIPAA-compliant Zoom videoconferencing. If participants are unable to join by Zoom videoconferencing, telephone (a format widely used in Cognitive Behavior Therapy (CBT) for Post Traumatic Stress Disorder (PTSD) treatment delivery and in CBT for depression) will be utilized. Ethical guidelines for providing telehealth over videoconferencing or phone will be followed.
  Arms: Treatment

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an internet- assisted Career-Oriented Work-Related Soft-skills Training (iCareer) intervention, infused with cognitive behavioral therapy, targeting individuals ages 16-24 with mental health conditions, to improve employment outcomes. The overall objective is to help transition-age youth (TAY) with psychiatric disabilities achieve optimal employment outcomes as part of successful transition to adulthood. Findings will have implications for enhancing and developing pre-employment services for TAY with psychiatric disabilities.

DETAILED DESCRIPTION:
The investigators propose to perform an open trial research study directed toward producing new knowledge about the Direct Skills Teaching intervention for employment related interpersonal "soft" skills. Soft skills are generally defined as social, emotional, interpersonal, adaptive, and problem-solving skills (Grugulis et al., 2009). The investigators will examine the feasibility of integrated Direct Skills Training modules in social, emotional, interpersonal, adaptive, and problem-solving skills (Soft Skills at Work (SSW)) on improving employment participation and success among transition age youth and young adults (TAY) with disabilities ages 18-24.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 16 and 24 years
2. Must speak English fluently
3. Receiving Individualized Education Program (IEP)/504 Plan or disability services within the past 24 months with primary disability types of psychiatric disability
4. No hospitalizations or suicide attempts within the past 2 months
5. Willing to provide informed consent (if younger than 18, parental consent) to participate in the study
6. Interested in improving work-related social skills

Exclusion Criteria:

1. Current presence of neurological disease or brain injury
2. Psychiatric instability such as gross psychosis or acute suicidality
3. Current alcohol or substance dependence
4. Hospitalization or suicide attempts in the past 2 months

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Higher Rates of Employment | 12 months post intervention
  Participants in iCareer will have higher rates of employment than participants in TAU alone as evidenced by self-report of acquiring a job.
Higher Number of Hours Worked | 12 months post intervention
  Participants in iCareer will have higher numbers hours worked than particiapants in TAU alone as evidenced by self-report of hours worked.
Increased Wages Earned | 12 months post intervention
  Participants in iCareer will have higher wages earned than participants in TAU alone as evidenced by self-report of wages earned.
Improved Job Related Social Skills | 12 months post intervention
  Participants in iCareer will have better job-related social skills than in TAU alone as evidenced by higher scores on the Job Related Social Skills Checklist (Reganick, 1995).

SECONDARY OUTCOMES:
Reduced Depressive Symptoms | 12 months post intervention
  Participants in iCareer will report less depression and overall symptoms than participants in TAU services alone as evidenced by lower scores on the Patient Health Questionnaire-9 (PHQ-9; Kroeneke et al., 2001)
Improved Functional Status | 12 months post intervention
  Participants in iCareer will report improved functional status related to their disability than participants in TAU alone as evidenced by lower scores on the Sheehan Disability Scale (Sheehan,1983) and lower scores on the BASIS-32 (Eisen et al., 1994).
Reduced Mental Illness Stigma | 12 months post intervention
  Participants in iCareer will report less stigma related to mental illness than participants in TAU alone as evidenced by lower scores on the Brief Version of the Internalized Stigma of Mental Illness Scale (ISMI-10; Boyd et al., 2014).
Increased Work Empowerment | 12 months post intervention
  Participants in iCareer will report increased work empowerment compared to participants in TAU services alone as evidenced by higher scores on the Work Related Self-Efficacy Scale (WSS; Waghorn et al., 2005).
Increased Job Satisfaction | 12 months post intervention
  Participants in iCareer will report increased job satisfaction compared to participants in TAU services alone as evidenced by higher scores on the Occupational Self-Efficacy Scale- Short Form (OSES; Schyns & von Collani, 2002).
Increased Job Motivation | 12 months post intervention
  Participants in iCareer will report increased motivation to get employment compared to participants in TAU services alone as evidenced by lower scores on the Perceived Employment Barriers Survey (PEBS; Hong et al., 2014) and higher scores on the Short Employment Hope Scale (Hong &Choi, 2013).

CONTACTS AND LOCATIONS:
Overall Officials: Weili Lu, PhD, Principal Investigator — Rutgers University, School of Health Professions
Locations (1):
- Rutgers Univeristy, Newark- Office of Disability Services, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Secondary use of data may be available to researchers after the completion of the study, provided through de-identified data deposited to the data repository, Interuniversity Consortium for Political and Social Research (ICPSR) as part of the grant award agreement required by the funding agency, the National Institute on Disability, Independent Living, and Rehabilitation Research (NIDILRR). The ICPSR will further ensure that the data will in no way contain any identifying information for participants.
Time Frame: Secondary use of data may be available to researchers after the completion of the study, provided through de-identified data deposited to the data repository, Interuniversity Consortium for Political and Social Research (ICPSR) as part of the grant award agreement required by the funding agency, the National Institute on Disability, Independent Living, and Rehabilitation Research (NIDILRR). The ICPSR will further ensure that the data will in no way contain any identifying information for participants.
Access Criteria: Secondary use of data may be available to researchers after the completion of the study, provided through de-identified data deposited to the data repository, Interuniversity Consortium for Political and Social Research (ICPSR) as part of the grant award agreement required by the funding agency, the National Institute on Disability, Independent Living, and Rehabilitation Research (NIDILRR). The ICPSR will further ensure that the data will in no way contain any identifying information for participants.